CLINICAL TRIAL: NCT06796803
Title: Camrelizumab and Rivoceranib Plus HAIC As Conversion Therapy for Potentially Resectable Intermediate-advanced Hepatocellular Carcinoma: a Multicenter, Open-label, Randomized, Phase 2/3 Study
Brief Title: Camrelizumab Combined with Rivoceranib and Hepatic Arterial Infusion Chemotherapy (HAIC) As Conversion Therapy for Potentially Resectable Hepatocellular Carcinoma(HCC)
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-HCC-II/III-026; 2024ZD0520401 (Other Grant/Funding Number: National Health Commission of the people's Republic of China)
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Potentially Resectable Hepatocellular Carcinoma
Keywords: conversion therapy; hepatocellular carcinoma; camrelizumab and rivoceranib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- camrelizumab + rivoceranib + HAIC (Experimental)
  Interventions: Drug: camrelizumab combined with rivoceranib and HAIC
- camrelizumab + rivoceranib (Active Comparator)
  Interventions: Drug: camerlizumab + rivoceranib

INTERVENTIONS:
Drug: camrelizumab combined with rivoceranib and HAIC — systemic therapy combined with locoregional theraphy as conversion therapy
  Arms: camrelizumab + rivoceranib + HAIC
Drug: camerlizumab + rivoceranib — systemic therapy
  Arms: camrelizumab + rivoceranib

SUMMARY:
The purpose of this phase 2/3 study is to investigate the efficacy and safety of camrelizumab combined with rivoceranib and hepatic arterial infusion chemotherapy (HAIC) as conversion therapy for Potentially Resectable HCC.

DETAILED DESCRIPTION:
This is a multicenter, open-label, randomized study designed to evaluate the efficacy and safety of camrelizumab combined with rivoceranib and HAIC as conversion therapy.

Eligible patients will be randomized into camrelizumab + rivoceranib + HAIC group and camrelizumab + rivoceranib group. Patients in camrelizumab + rivoceranib + HAIC group will receive systemic therapy and no more than 6 cycles HAIC procedure. Tumor response assessment using CT and/or MRI will be conducted according to RECIST v1.1. Those who are assessed as CR/PR or SD and considered suitable for curative hepatic resection will receive surgry. Surgical approaches will be tailored to the individual patient according to local standards with the goal of achieving R0 resection.The first administration of postoperative camrelizumab + rivoceranib treatment is recommended to start within 4-6 weeks after surgery, requiring full recovery from the surgery prior to post-operative camrelizumab + rivoceranib treatment. Patients in camrelizumab + rivoceranib group will receive the systemic therapy until progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form (ICF)
2. Aged ≥18 years and ≤75 years at time of signing ICF
3. Documented diagnosis of HCC confirmed by histology/cytology or clinically
4. Patients with BCLC stage B (the sum of number of tumors and the maximum diameter of the largest tumor exceeding Up-to-7 criteria) and BCLC stage C without extrahepatic metastasis: ① tumors confined to one lobe (left, right, or middle lobe), or tumors in one lobe are present alongside a single tumor with diameter ≤5 cm or up to three tumors each with diameter ≤3 cm in the remaining lobes; ②No PVTT involving the contralateral liver lobe or reaching the superior mesenteric vein. And no tumor thrombus of the inferior vena cava reaching right atrium
5. At least one measurable lesion (per RECIST v1.1) untreated lesion
6. ECOG performance status of 0 or 1
7. Child-Pugh ≤7 score
8. Life expectancy ≥12 weeks
9. Adequate organ function
10. No prior anti-tumor systemic therapies for HCC

Exclusion Criteria:

1. Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
2. Other active malignant tumor except HCC within 5 years or simultaneously
3. Prior locoregional therapy (such as TACE、TAE、HAIC、TARE)
4. There is an absolute contraindication to HAIC
5. History of hepatic encephalopathy
6. Diffuse HCC, intrahepatic tumor burden > 50%
7. PVTT reaching the superior mesenteric vein, and bilateral PVTT are present
8. Clinically significant ascites
9. Prior allogeneic stem cell or solid organ transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2028-02-20 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
R0 rate | 24 months
  R0 rate defined as the proportion of patients who accomplish the complete resection of tumor with pathologically confirmed negative margin
OS | 24 months
  Overall survival (OS) after randomization, defined as the time from randomization to death from any cause

SECONDARY OUTCOMES:
EFS | 24 months
  Event-free survival (EFS), defined as the time from randomization to progression (RECIST v1.1), recurrence and death from any cause
ORR | 24 months
  Objective response rate (ORR), defined as the percentage of subjects with complete response (CR) or partial response (PR) evaluated based on RECIST v1.1. CR: disappearance of all target lesions. PR: At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. Overall Response (OR)=CR+PR.
DCR | 24 months
  Disease Control Rate (DCR), defined as the percentage of subjects with complete response, partial response or stable disease (SD) ≥ 8 weeks evaluated based on RECIST v1.1. Complete response (CR) was defined as Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response (PR) was defined as at least a 30% decrease in the sum of the diameter of TL, taking as reference the baseline sum of diameters. Stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
pCR rate | 24 months
  Pathological complete regression (pCR) rate, defined as the proportion of patients with no evidence of vital residual tumor cells on the complete resected specimen. pCR status will be analyzed by local pathologists at each site
MPR rate | 24 months
  MPR rate, defined as the proportion of patients with evidence of vital residual tumor cells <50% on the resected specimen. MPR status will be analyzed by local pathologists at each site
AE | 24 months
  Adverse events are graded according to the NCI-CTCAE (Version 5.0)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided